CLINICAL TRIAL: NCT01848080
Title: A Tai Chi Based Exercise Program Provided Via Telerehabilitation Compared to During Home Visits in Persons Post-Stroke Who Have Returned Home Without Intensive Rehabilitation: A Randomized, Non-inferiority Clinical Trial
Brief Title: A Randomized, Non-inferiority Clinical Trial of CVA Telerehabilitation Treatments - TelePhysioTaiChi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Université de Montréal (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Michel Tousignant, Professor, PH.D., Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-217-S1
Record Dates: First submitted 2013-04-26; First posted 2013-05-07 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Stroke
Keywords: Telemedicine; Telerehabilitation; Acute Stroke; Tai Chi; Tai Ji; Rehabilitation; Home care services; Single blind method; Randomized controlled trial
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai chi program via Telerehabilitation (Experimental): An individualized exercise program, based on Tai Chi, was developed by our team for previous studies aiming to improve balance in elderly, diabetic individuals and in frail, elderly individuals with balance problems. The exercise program consists of movements based on a combination of alignments and body-specific orientations, weight transfers and changes in direction inspired by Tai Chi. This group will receive this program via telerehabilitation.
  Interventions: Behavioral: Tai Chi based exercise program
- Tai chi program via home visits (Active Comparator): An individualized exercise program, based on Tai Chi, was developed by our team for previous studies aiming to improve balance in elderly, diabetic individuals and in frail, elderly individuals with balance problems. The exercise program consists of movements based on a combination of alignments and body-specific orientations, weight transfers and changes in direction inspired by Tai Chi. This group will receive this program via home visits.
  Interventions: Behavioral: Tai Chi based exercise program

INTERVENTIONS:
Behavioral: Tai Chi based exercise program — A Tai Chi based exercise program that uses movement repetition favoring directional adjustments in space, supervised by a physiotherapist, has been shown to be effective in improving balance in individuals with physical impairments, including those presenting with sequelae following a stroke.

SUMMARY:
Telerehabilitation is a promising alternative approach that can help improve access to rehabilitation services once patients are discharged home after stroke. The investigators therefore postulate a non-inferiority hypothesis of the telerehabilitation approach compared to home visits to improve balance problem related to stroke. The platform used will be based on a technological infrastructure that was developed and tested in previous telerehabilitation studies. The study is a randomized control trial (RCT).The study population of interest will target individuals who have had a stroke who stayed in a hospital or chronic stroke population. Participants will be recruited during the hospitalization period at each of the three sites or in the community. The investigators expect to recruit 240 participants, 120 per group. The first evaluation will be conducted at recruitment to establish the baseline measures. The two other evaluations will be conducted 2 months (T2) and four months (T3) following recruitment.

ELIGIBILITY:
Inclusion Criteria:

* have had a stroke with a Rankin score of 2 or 3;
* was not referred to an Intensive Functional Rehabilitation Unit (IFRU) and returned home following discharge from hospital;
* understands instructions to allow participation in evaluations and interventions;
* has a balance problem as evidenced by a score between 46 and 54 on the Berg Balance Scale96;
* has a caregiver that would be available during the telerehabilitation sessions to ensure safety during exercises;
* live in an area serviced by high speed Internet.

Exclusion Criteria:

* severe body hemineglect;
* significant hemianopsia visual problems accompanied by hemineglect;
* uncontrolled medical problems;
* moderate to severe aphasia

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mobility at 2 and 4 months | before the intervention, month 2 and month 4
  Community balance and mobility Scale.
Change from baseline in Balance at 2 and 4 months | before the intervention, month 2 and month 4
  Community balance and mobility Scale.

SECONDARY OUTCOMES:
Change from baseline walking speed at 2 and 4 months | before the intervention, month 2, month 4
  Speed: Timed up and go (TUG),
Change from baseline Psychological Attitudes related to balance at 2 and 4 months | before the intervention, month 2, month 4
  Self efficacy: General Perceived Self efficacy
Change from baseline Quality of life at 2 and 4 month | before the intervention, month 2, month 4
  Quality of life: Reintegration ti normal Living Index (RNLI)
Change from Baseline Satisfaction with the care received at 2 and 4 months | before the intervention, month 2, month 4
  Satisfaction with the care received = Health care satisfaction questionnaire
Change from Baseline Cost of services from the perspective of the health system at 2 and 4 months | before the intervention, month 2, month 4
  Cost of services from the perspective of the health system = "Cost-analysis of telemedicine" from the Minnesota University
Change from baseline walking endurance at 2 and 4 months | before the intervention, month 2 and month 4
  distance in meters walked two minutes
Change from baseline aptitude for Balance at 2 and 4 months | before the intervention, month 2 and month 4
  Four-Squares Test
Change from baseline Strength of lower limbs at 2 and 4 months | before the intervention, month 2 and month 4
  Sit to Stand Test
Change from baseline Psychological Attitudes related to mobility at 2 and 4 months | before the intervention, month 2, month 4
  fear of falling: Activities-specific Balance confidence scale

CONTACTS AND LOCATIONS:
Overall Officials: Michel Tousignant, PhD, Principal Investigator — Research Centre on Aging
Locations (3):
- Canada (3):
  - Hôpital Charles-LeMoyne, Longueuil
  - Centre de recherche interdisciplinaire en réadaptation du Montréal métropolitain, Montreal
  - Research Centre on Aging, Sherbrooke

REFERENCES:
- [Background] Tousignant M, Corriveau H, Kairy D, Berg K, Dubois MF, Gosselin S, Swartz RH, Boulanger JM, Danells C. Tai Chi-based exercise program provided via telerehabilitation compared to home visits in a post-stroke population who have returned home without intensive rehabilitation: study protocol for a randomized, non-inferiority clinical trial. Trials. 2014 Jan 30;15:42. doi: 10.1186/1745-6215-15-42. PMID 24479760
- See also: Complete and published research protocol — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3912257/pdf/1745-6215-15-42.pdf